CLINICAL TRIAL: NCT04394988
Title: Total 102 Natural Orifice Specimen Extractions Following Laparoscopic Colorectal Resections
Status: Completed | Type: Observational
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Ersin Gündoğan, Doctor- lecturer-Principal Investigator, Inonu University
Other Study IDs: 2018/21-41
Record Dates: First submitted 2020-05-15; First posted 2020-05-20 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Incisional Hernia; Incision Infection
Keywords: natural orifice surgery; minimally invasive surgery; colon cancer; laparoscopic colorectal
MeSH Terms: conditions — Incisional Hernia; Surgical Wound Infection; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In the development of surgical technique, laparoscopic surgery has created a major breaking point. Although laparoscopy (decreased hospital stay, decreased incisional hernia and wound infection rate…) provides a remarkable advantage compared to open surgery, the need for the extraction site incision could not bring the incision-related morbidity rates to the desired level. That's why SILS and natural hole surgery came to the fore. Colorectal surgery was also affected by this process, and the laparoscopic colectomy procedure combined with transrectal colon extraction was first performed in 1993 (1). Although its use increased gradually after this period, it could not reach the expected levels and this could not resolve the concerns on natural hole surgery.

In this article, our aim is to present the single center results of the patients who performed the extraction with the NOSE method after laparoscopic colorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent laparoscopic - natural orifice colectomy.

Exclusion Criteria:

* patients with missing data
* patients who underwent open colectomy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients who underwent laparoscopic-natural orifice colectomy at General Surgery Clinic in Inonu University between January 2013 and July 2018
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
complications due to incision and aesthetic score | 6 months
  Hernia, infection, hospital stay and aesthetic score

CONTACTS AND LOCATIONS:
Overall Officials: Ersin Gundogan, MD, Principal Investigator — Inonu University
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gundogan E, Aktas A, Kayaalp C, Gonultas F, Sumer F. Two cases of laparoscopic total colectomy with natural orifice specimen extraction and review of the literature. Wideochir Inne Tech Maloinwazyjne. 2017 Sep;12(3):291-296. doi: 10.5114/wiitm.2017.69227. Epub 2017 Jul 27. PMID 29062451
- [Background] Kayaalp C, Kutluturk K, Yagci MA, Ates M. Laparoscopic right-sided colonic resection with transluminal colonoscopic specimen extraction. World J Gastrointest Endosc. 2015 Sep 10;7(12):1078-82. doi: 10.4253/wjge.v7.i12.1078. PMID 26380054
- [Background] Karagul S, Kayaalp C, Sumer F, Ertugrul I, Kirmizi S, Tardu A, Yagci MA. Success rate of natural orifice specimen extraction after laparoscopic colorectal resections. Tech Coloproctol. 2017 Apr;21(4):295-300. doi: 10.1007/s10151-017-1611-2. Epub 2017 Apr 26. PMID 28447167
- [Background] Awad ZT, Griffin R. Laparoscopic right hemicolectomy: a comparison of natural orifice versus transabdominal specimen extraction. Surg Endosc. 2014 Oct;28(10):2871-6. doi: 10.1007/s00464-014-3540-8. Epub 2014 May 2. PMID 24789131
- [Derived] Gundogan E, Kayaalp C, Alinak Gundogan G, Sumer F. Total 102 natural orifice specimen extraction following laparoscopic colorectal resections. Updates Surg. 2023 Jan;75(1):197-203. doi: 10.1007/s13304-022-01412-4. Epub 2022 Nov 1. PMID 36319790